CLINICAL TRIAL: NCT04943289
Title: Phase IA Trial of Intrathecal Administration of Human Umbilical Cord Blood-Derived Cell Therapy (DUOC-01) in Adults With Primary Progressive Multiple Sclerosis (PPMS)
Brief Title: Intrathecal Administration of DUOC-01 in Adults With Primary Progressive Multiple Sclerosis
Acronym: DUOC for MS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00107012
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Primary Progressive Multiple Sclerosis
Keywords: Multiple Sclerosis, MS
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DUOC-01 (Experimental): Intrathecal Infusion of DUOC-01 and hydrocortisone. Cohort 1: 10 million cells Cohort 2: greater than 10 to 25 million cells Cohort 3: greater than 25 to 50 million cells
  Interventions: Biological: DUOC-01

INTERVENTIONS:
Biological: DUOC-01 — DUOC-01 is a population of cells expanded from donor human umbilical cord blood mononuclear cells. DUOC-01 cells are derived from CB CD14+ monocytes. DUOC-01 will be administered along with hydrocortisone via intrathecal injection.

SUMMARY:
This study is a prospective Phase 1a open-label single- center trial. It will assess the safety of intrathecal administration of DUOC-01 cells to adults with Primary Progressive Multiple Sclerosis (PPMS). DUOC-01 is a population of cells expanded from donated human umbilical cord blood cells and is intended for treatment of neurodegenerative and demyelinating diseases. There will be approximately 20 participants enrolled. Exploratory objectives include changes in MS assessment scores, changes in brain MRI findings, and changes in blood biomarkers.

DETAILED DESCRIPTION:
This study is a prospective phase 1a open-label, single center trial. It is designed to assess the safety of administration of escalating doses of DUOC-01 intrathecally to adults with PPMS. DUOC-01 is a population of cells expanded from donated human umbilical cord blood mononuclear cells. Immunodepletion and selection studies demonstrated that DUOC-01 cells are derived from CB CD14+ monocytes. Based on pre-clinical rodent models, this cell product is considered a candidate for the treatment of injury-induced Central Nervous System (CNS) demyelination and modulation of neuroinflammation.

Approximately 20 participants will be enrolled. DUOC-01 will be infused into the cerebrospinal fluid (intrathecal infusion). The first 3 subjects will receive a single dose of 10 million cells (cohort 1). The next 3 subjects will receive a single intrathecal dose of >10 to 25 million cells (cohort 2), if manufacturing of this yield is reliable. The final 14 patients will receive a single intrathecal dose of >25 to 50 million cells (cohort 3), if manufacturing of this yield is reliable. Subjects will be followed for 12 months post administration.

Participants will be identified and screened for eligibility for the study. HLA typing will be performed on the participant, and once results become available, several >4/6 matched cord blood units (CBUs) will be selected from the Carolinas Cord Blood Bank (CCBB), an FDA licensed public cord blood bank at Duke University in Durham, NC. Cord blood units will have complete donor screening and testing per banking regulations.

The frozen CBU will be transferred to the GMP manufacturing facility at Duke University Medical Center per standard practice. Production, testing and release of DUOC-01 will take 19-21 days. Within 14 days prior to planned administration, subjects will receive a baseline brain MRI and be re-screened on MS assessments. Subjects will not be infused with DUOC-01 cells if they no longer meet inclusion criteria or if no qualifying DUOC-01 cells are available. If there is a failure of DUOC-01 manufacturing, a second cord blood unit, if available, will be utilized for repeat manufacturing.

DUOC-01 administration will occur by a trained clinician. A lumbar puncture (insertion of a needle into the lower back, into the cerebrospinal spinal fluid (CSF)) will be performed and baseline CSF samples will be obtained. The DUOC-01 product will be injected into the CSF (intrathecally) and appropriate monitoring will be performed.

Post administration, all subjects will remain in the hospital for 24-hour observation. At 2 weeks post administration subjects will participate in a virtual visit to evaluate for adverse events. Subjects will receive follow up visits with functional evaluation, biomarker sampling and brain MRI at 3, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects must be 18-65 years of age
2. Diagnosis of primary progressive MS according to 2017 revised McDonald criteria (26)
3. EDSS score at screening 3.0-6.5 that was not acquired within the last 6 months
4. Stable disease state as evidenced by no significant change in EDSS (1 point or more) in the last 3 months
5. Patients must have a suitably matched, banked UCB per section 5.3
6. Able to complete a written informed consent prior to any study assessments
7. Patients of childbearing potential must practice effective contraception during the study, and be willing to continue contraception for at least 6 months after DUOC-01 dosing so that, in the opinion of the Investigator, they will not become pregnant during the course of the study.
8. Patient is a good candidate for the trial, in the opinion of the Investigators
9. Subjects on disease-modifying therapies upon entering the study must continue on these therapies as a concomitant treatment throughout the course of the study to minimize additional variables. However, changes in these disease-modifying therapies can occur at the clinician's discretion, if there are clinical reasons to do so, which would be documented.

Exclusion Criteria:

* 1. Prior organ, tissue, or stem cell transplant or cell therapy within 3 years of study entry 2. Diagnosis of a progressive neurological disorder other than MS 3. Active, chronic disease of the immune system other than MS 4. Any medical condition that the investigator deems as unsuitable with therapy 5. Inability to have an MRI brain scan, or lumbar puncture (i.e., claustrophobia, allergy to contrast, bleeding disorder, or on anticoagulation) 6. Intractable seizures 7. Chronic aspiration 8. Bleeding disorder 9. Evidence of HIV infection or HIV positive serology 10. Uncontrolled bacterial, viral, or fungal infection within 2 weeks of DUOC-01 administration, as defined by progression while on appropriate treatment 11. History of malignancy of any organ system within the past two years with the exception of basal cell carcinoma or squamous cell carcinoma of the skin that has been excised with clear margins. 12. Requirement of ventilatory support 13. Pregnant or breastfeeding or intention to become pregnant during the study 14. Active concurrent malignancy, or receiving concurrent radiotherapy, immunosuppressive medications for conditions other than MS, or cytotoxic chemotherapy 15. Patients with Suicidal Ideation in the past 6 months per screening on C-SSRS; patients with Suicidal Behavior in the past 2 years, except for Non-suicidal self-injurious behavior 16. Abnormal lab values:
* Total bilirubin>2.0 mg/dl unless due to Gilbert's syndrome
* AST or ALT > 5 times the ULN
* WBC <2.0x 103/μL
* ALC <0.5 x 103/ μL
* Serum creatinine >2x ULN
* eGFR <60 mg/mmol
* CD4 count <200 cells/mm3

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Incidence of IT administration adverse events | 2 weeks post infusion
  Total number of adverse events associated with DUOC-01 infusion
Incidence of adverse events attributed to the investigational product | 1 year post infusion
  Cumulative summary of adverse events related to DUOC-01

CONTACTS AND LOCATIONS:
Overall Officials: Beth Shaz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtzberg J, Buntz S, Gentry T, Noeldner P, Ozamiz A, Rusche B, Storms RW, Wollish A, Wenger DA, Balber AE. Reprint of: Preclinical characterization of DUOC-01, a cell therapy product derived from banked umbilical cord blood for use as an adjuvant to umbilical cord blood transplantation for treatment of inherited metabolic diseases. Cytotherapy. 2015 Sep;17(9):1314-26. doi: 10.1016/j.jcyt.2015.07.014. PMID 26276011
- [Background] Saha A, Buntz S, Scotland P, Xu L, Noeldner P, Patel S, Wollish A, Gunaratne A, Gentry T, Troy J, Matsushima GK, Kurtzberg J, Balber AE. A cord blood monocyte-derived cell therapy product accelerates brain remyelination. JCI Insight. 2016 Aug 18;1(13):e86667. doi: 10.1172/jci.insight.86667. PMID 27699230
- [Background] Tracy ET, Zhang CY, Gentry T, Shoulars KW, Kurtzberg J. Isolation and expansion of oligodendrocyte progenitor cells from cryopreserved human umbilical cord blood. Cytotherapy. 2011 Jul;13(6):722-9. doi: 10.3109/14653249.2011.553592. Epub 2011 Feb 22. PMID 21341973
- [Background] Tracy E, Aldrink J, Panosian J, Beam D, Thacker J, Reese M, Kurtzberg J. Isolation of oligodendrocyte-like cells from human umbilical cord blood. Cytotherapy. 2008;10(5):518-25. doi: 10.1080/14653240802154586. PMID 18608351
- [Background] Scotland P, Buntz S, Noeldner P, Saha A, Gentry T, Kurtzberg J, Balber AE. Gene products promoting remyelination are up-regulated in a cell therapy product manufactured from banked human cord blood. Cytotherapy. 2017 Jun;19(6):771-782. doi: 10.1016/j.jcyt.2017.03.004. Epub 2017 Apr 5. PMID 28391986
- [Background] Kurtzberg J, Buntz S, Gentry T, Noeldner P, Ozamiz A, Rusche B, Storms RW, Wollish A, Wenger DA, Balber AE. Preclinical characterization of DUOC-01, a cell therapy product derived from banked umbilical cord blood for use as an adjuvant to umbilical cord blood transplantation for treatment of inherited metabolic diseases. Cytotherapy. 2015 Jun;17(6):803-815. doi: 10.1016/j.jcyt.2015.02.006. Epub 2015 Mar 12. PMID 25770677